CLINICAL TRIAL: NCT01594229
Title: A Phase 1 Study Evaluating the Safety and Pharmacokinetics of ABT-199 in Combination With Bendamustine/Rituximab (BR) in Subjects With Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: A Study Evaluating the Safety and Pharmacokinetics of ABT-199 in Combination With Bendamustine/Rituximab (BR) in Subjects With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-630
Record Dates: First submitted 2012-04-20; First posted 2012-05-09 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Pharmacokinetics; Maximum Tolerated Dose; Safety; Bendamustine; Non-Hodgkin's Lymphoma; Rituximab; ABT-199; Cancer; Preliminary Efficacy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms | interventions — venetoclax; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Non-Hodgkin's Lymphoma (NHL)
  Interventions: Drug: ABT-199; Drug: Rituximab; Drug: Bendamustine

INTERVENTIONS:
Drug: ABT-199 — ABT-199 is taken orally once daily for 3 days out of each 28 day cycle. This is a dose escalation study, therefore the dose of ABT-199 will change throughout the study.
Drug: Rituximab — Rituximab will be given by intravenous infusion for 1 day out of each 28 day cycle.
Drug: Bendamustine — Bendamustine will be given by intravenous infusion for 2 days out of each 28 day cycle.

SUMMARY:
This is a Phase 1, open-label, multicenter study evaluating the safety, pharmacokinetic profile, and preliminary efficacy of ABT-199 in combination with Bendamustine/Rituximab in approximately 60 subjects with relapsed or refractory non-Hodgkin's lymphoma. This study will evaluate the safety and pharmacokinetic profile of ABT-199 in approximately 60 subjects when administered in combination with Bendamustine/Rituximab following a dose escalation scheme, with the objective of defining the dose limiting toxicity and the maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have histologically documented diagnosis of non-Hodgkin's lymphoma as defined by a B-cell neoplasm in the World Health Organization classification scheme except as noted in exclusion criteria.
* Subject (non-diffuse large B-cell lymphoma) must have relapsed or refractory non-Hodgkin's lymphoma, and require treatment in the opinion of the investigator.
* Subject with diffuse large B-cell lymphoma must have relapsed diffuse large B-cell lymphoma or must have progressed after salvage therapy (with or without standard chemotherapy) for diffuse large B-cell lymphoma. The subject must have received first line therapy with Rituximab-Cyclophosphamide, Hydroxydaunomycin, Vincristine (Oncovin), Prednisone (R-CHOP) [or a similar standard rituximab-containing front-line chemoimmunotherapy regimen including, but not limited to Etoposide, Prednisone, Vincristine (Oncovin), Cyclophosphamide, Doxorubicin (Hydrochloride) + Rituximab (EPOCH + R); Rituximab, Cyclophosphamide, Etoposide, Procarbazine, Prednisone (RCEPP); Rituximab, Cyclophosphamide, Mitoxantrone (Novantrone), Vincristine (Oncovin), Prednisone (RCNOP); Dose-adjusted-Etoposide, Prednisone, Vincristine(Oncovin), Cyclophosphamide, Doxorubicin (Hydrocloride) (DA-EPOCH); and Rituximab, Cyclophosphamide, Etoposide, Vincristine (Oncovin), Prednisone (RCEOP)].
* Subject must have adequate coagulation, renal, and hepatic function, per laboratory reference range at Screening.

Exclusion Criteria:

* Subject has been diagnosed with Post-Transplant Lymphoproliferative Disease, Burkitt's lymphoma, Burkitt-like lymphoma, lymphoblastic lymphoma/leukemia, chronic lymphocytic leukemia, small lymphocytic lymphoma or mantle cell lymphoma (MCL).
* Subject has refractory diffuse large B-cell lymphoma, defined as meeting any of the following criteria:

  * Subject progressed during or within 3 months of completion of a planned course of first-line therapy with Rituximab-Cyclophosphamide, Hydroxydaunomycin, Vincristine (Oncovin), Prednisone (R-CHOP) or an equivalent regimen;
  * Subject had no response (i.e., stable disease only) to first-line therapy with R-Cyclophosphamide, Hydroxydaunomycin, Vincristine (Oncovin), Prednisone (R-CHOP) or an equivalent regimen;
  * Subject progressed during or within 2 months of completion of their last planned course of salvage therapy with chemotherapy (with or without rituximab, may include autologous stem cell transplant).
* Subject has tested positive for human immunodeficiency virus (HIV).
* Subject has a cardiovascular disability status of New York Heart Association Class greater or equal to 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity, results in fatigue, palpitations, dyspnea or anginal pain.
* Subject has a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease that in the opinion of the Investigator would adversely affect his/her participating in this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose of ABT-199 when administered with Bendamustine and Rituximab in subjects with relapsed or refractory non-Hodgkin's lymphoma | 3 days of study drug administration within the 28-day cycle at the designated cohort dose
  Protocol-defined events, which can not be attributed by the investigator to a clearly identifiable cause such as tumor progression, concurrent illness, or concomitant medication, will be considered a dose limiting toxicity
Determination of peak concentration (Cmax), trough concentration (Ctrough) and/or area under the concentration versus time curve (AUC) of ABT-199, Bendamustine and Rituximab in the dose escalation cohort | Up to Cycle 6 for ABT-199 and Bendamustine, Up to Cycle 11 for Rituximab
  Protocol-defined events, which can not be attributed by the investigator to a clearly identifiable cause such as tumor progression, concurrent illness, or concomitant medication, will be considered a dose limiting toxicity
Number of participants with adverse events as a measure of safety and tolerability | First 5 days of study drug administration, weekly through Cycle 2 and then Day 1 of each Cycle for an anticipated maximum duration of 6 months
  Adverse event monitoring, vital signs, physical examination, lymphocyte enumeration, 12-lead ECG, 2D echocardiogram/multiple gated acquisition scan (MUGA), and laboratory assessments
Determination of the recommended Phase 2 dose of ABT-199 when administered with Bendamustine and Rituximab in subjects with relapsed or refractory non-Hodgkin's lymphoma | 3 days of study drug administration within the 28-day cycle at the designated cohort dose
  Protocol-defined events, which can not be attributed by the investigator to a clearly identifiable cause such as tumor progression, concurrent illness, or concomitant medication, will be considered a dose limiting toxicity

SECONDARY OUTCOMES:
Evaluate preliminary data regarding progression-free survival when ABT-199 is administered in combination with Bendamustine and Rituximab | Tumor Assessments: Approximately every 2 cycles through Cycle 17 then every 6 cycles thereafter; Clinical Disease Assessment: Weekly through Cycle 2, then every cycle thereafter
  Tumor response or clinical disease progression
Evaluate preliminary data regarding overall survival and duration of overall response when ABT-199 is administered in combination with Bendamustine and Rituximab. | Tumor Assessments: Approximately every 2 cycles through Cycle 17 then every 6 cycles thereafter; Clinical Disease Assessment: Weekly through Cycle 2, then every cycle thereafter
  Tumor response or clinical disease progression
Evaluate preliminary data regarding objective response rate when ABT-199 is administered in combination with Bendamustine and Rituximab | Tumor Assessments: Approximately every 2 cycles through Cycle 17 then every 6 cycles thereafter; Clinical Disease Assessment: Weekly through Cycle 2, then every cycle thereafter
  Tumor response or clinical disease progression
Evaluate preliminary data regarding time to tumor progression when ABT-199 is administered in combination with Bendamustine and Rituximab. | Tumor Assessments: Approximately every 2 cycles through Cycle 17 then every 6 cycles thereafter; Clinical Disease Assessment: Weekly through Cycle 2, then every cycle thereafter
  Tumor response or clinical disease progression

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (8):
- United States (8):
  - Ucsd /Id# 67350, La Jolla, California
  - University of California, Los Angeles /ID# 67343, Los Angeles, California
  - Emory University Hospital /ID# 67349, Atlanta, Georgia
  - Georgia Regents University /ID# 67342, Augusta, Georgia
  - Ingalls Memorial Hosp /ID# 67344, Harvey, Illinois
  - Johns Hopkins University /ID# 67345, Baltimore, Maryland
  - Henry Ford Health System /ID# 67346, Detroit, Michigan
  - University of Texas MD Anderson Cancer Center /ID# 69222, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Vos S, Swinnen LJ, Wang D, Reid E, Fowler N, Cordero J, Dunbar M, Enschede SH, Nolan C, Petrich AM, Ross JA, Salem AH, Verdugo M, Agarwal S, Zhou L, Kozloff M, Nastoupil LJ, Flowers CR. Venetoclax, bendamustine, and rituximab in patients with relapsed or refractory NHL: a phase Ib dose-finding study. Ann Oncol. 2018 Sep 1;29(9):1932-1938. doi: 10.1093/annonc/mdy256. PMID 30060083